CLINICAL TRIAL: NCT07184060
Title: A Prospective Observational Study on Pulmonary Hypertension in Patients With Obstructive Sleep Apnea: Correlation of Apnea-Hypopnea Severity With Pulmonary Artery Pressures
Brief Title: Echocardiographic Assessment of Pulmonary Hypertension in Obstructive Sleep Apnea
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ashraqat Tony Badawy, resident at the of Chest Diseases department, Assiut University
Other Study IDs: Pulmonary Hypertension in OSA
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Obstructive Sleep Apnea (OSA); Pulmonary Hypertension
Keywords: obstructive sleep apnea; pulmonary hypertension
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult patients with confirmed OSA: Eligible participants are 18-65 years old and diagnosed with OSA (AHI ≥ 5 events/hour) confirmed through full-night polysomnographic sleep study. Patients will be stratified into mild (AHI 5-14), moderate (AHI 15-29), and severe OSA (AHI ≥ 30). Exclusion criteria include patients with secondary PH (from cardiac causes, chronic thromboembolic disease, or pulmonary conditions), chronic vasodilator therapy, long-term oxygen therapy, advanced organ failure, neuromuscular or chest wall deformities, obesity hypoventilation syndrome, or malignancy. The expected sample size is 55 patients, ensuring enough statistical power to detect associations. Demographic, clinical, echocardiographic, radiological, and sleep study parameters will be collected for each patient.

SUMMARY:
This study investigates the association between obstructive sleep apnea (OSA) and pulmonary hypertension (PH), focusing on the relationship between OSA severity and pulmonary arterial pressures in adult patients.

DETAILED DESCRIPTION:
This prospective, observational, cross-sectional study will be conducted in the pulmonology and sleep medicine departments of Assiut University. Patients diagnosed with OSA through overnight polysomnography will be assessed for the presence and severity of PH using echocardiography. The study aims to determine whether OSA serves as an independent risk factor for PH and whether the severity of OSA, as measured by apnea-hypopnea index (AHI) and oxygen desaturation index (ODI), correlates with echocardiographic indicators of PH. Data will be analyzed using standardized statistical methods to establish links between OSA severity and hemodynamic changes.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-65 years

Diagnosed with obstructive sleep apnea (OSA) by full-night polysomnography

Apnea-Hypopnea Index (AHI) ≥ 5 events/hour

Exclusion Criteria:

Secondary pulmonary hypertension due to:Chronic pulmonary diseases, Left ventricular heart disease and Chronic thromboembolic disorders

Use of pulmonary vasodilator therapy

Long-term oxygen therapy (LTOT)

Respiratory neuromuscular weakness

Chest wall deformities

End-organ failure (cardiac, renal, hepatic)

Malignancy

Obesity hypoventilation syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants are 18-65 years old and diagnosed with OSA (AHI ≥ 5 events/hour) confirmed through full-night polysomnographic sleep study. Patients will be stratified into mild (AHI 5-14), moderate (AHI 15-29), and severe OSA (AHI ≥ 30). Exclusion criteria include patients with secondary PH (from cardiac causes, chronic thromboembolic disease, or pulmonary conditions), chronic vasodilator therapy, long-term oxygen therapy, advanced organ failure, neuromuscular or chest wall deformities, obesity hypoventilation syndrome, or malignancy. The expected sample size is 55 patients, ensuring enough statistical power to detect associations. Demographic, clinical, echocardiographic, radiological, and sleep study parameters will be collected for each patient.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Mean Pulmonary Artery Pressure | baseline
  The primary objective is to assess the presence and degree of pulmonary hypertension (measured by echocardiography) in OSA patients.

IPD SHARING:
Plan to Share IPD: No